CLINICAL TRIAL: NCT04291794
Title: Mean Arterial Pressure Reduction During the First Ten Minutes After General Anesthesia Induction Using Propofol Bolus or Tritiated Target-infusion: Superiority Randomized Controlled Trial
Brief Title: Mean Arterial Pressure Reduction Anesthesia Induction Using Propofol Bolus or Tritiated Target-infusion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brasilia University Hospital (Other)
Responsible Party: Principal Investigator, Gabriel Magalhaes Nunes Guimaraes, Voluntary professor, Brasilia University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: tccgui2019
Record Dates: First submitted 2020-02-26; First posted 2020-03-02 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Hypotension on Induction; Hypnotic Intoxication
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant and outcomes Assessor will not know group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional bolus induction (Active Comparator): Hypnotic component of general anesthesia induction will be a single bolus of propofol 2mg/kg followed by turning on sevoflurane 2% at a fresh gas flow of 2L/min.
  Interventions: Drug: Propofol
- Target-controlled induction (Experimental): Hypnotic component of general anesthesia induction will be target-controlled propofol infusion tritiated to loss of consciousness. Propofol target-controlled infusion will be maintained.
  Interventions: Drug: Propofol Injection [Diprivan]

INTERVENTIONS:
Drug: Propofol — 2mg/kg single bolus
  Arms: Conventional bolus induction
Drug: Propofol Injection [Diprivan] — Tritiated Target-Controlled Infusion
  Arms: Target-controlled induction

SUMMARY:
To compare haemodynamics and bispectral index values between conventional bolus propofol induction and target-controlled propofol infusion.

DETAILED DESCRIPTION:
To compare mean arterial pressure, heart rate and bispectral index values between conventional bolus propofol induction and target-controlled propofol infusion.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for general anesthesia;
* No contraindication for propofol.

Exclusion Criteria:

* Data loss;
* Protocol violation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2020-09-25 (Estimated); Study Completion 2020-11-27 (Estimated)

PRIMARY OUTCOMES:
Mean arterial pressure after 2 minutes | 2 minutes after general anesthesia induction
  Mean arterial pressure using non-invasive device
Mean arterial pressure after 4 minutes | 4 minutes after general anesthesia induction minutes after general anesthesia induction
  Mean arterial pressure using non-invasive device
Mean arterial pressure after 6 minutes | 6 minutes after general anesthesia induction minutes after general anesthesia induction
  Mean arterial pressure using non-invasive device
Mean arterial pressure after 8 minutes | 8 minutes after general anesthesia induction minutes after general anesthesia induction
  Mean arterial pressure using non-invasive device
Mean arterial pressure after 10 minutes | 10 minutes after general anesthesia induction minutes after general anesthesia induction
  Mean arterial pressure using non-invasive device

SECONDARY OUTCOMES:
Heart Rate after 2 minutes | 2 minutes after general anesthesia induction
  Heart rate (pulse rate) using non-invasive device.
Heart Rate after 4 minutes | 4 minutes after general anesthesia induction
  Heart rate (pulse rate) using non-invasive device.
Heart Rate after 6 minutes | 6 minutes after general anesthesia induction
  Heart rate (pulse rate) using non-invasive device.
Heart Rate after 8 minutes | 8 minutes after general anesthesia induction
  Heart rate (pulse rate) using non-invasive device.
Heart Rate after 10 minutes | 10 minutes after general anesthesia induction
  Heart rate (pulse rate) using non-invasive device.
Bispectral Index after 2 minutes | 2 minutes after general anesthesia induction
  Bispectral Index (BIS) using non-invasive device. At values near 100 mean patient is more likely to be awake and at values below 60 are more likely to be under general anesthesia.
Bispectral Index after 4 minutes | 4 minutes after general anesthesia induction
  Bispectral Index (BIS) using non-invasive device. At values near 100 mean patient is more likely to be awake and at values below 60 are more likely to be under general anesthesia.
Bispectral Index after 6 minutes | 6 minutes after general anesthesia induction
  Bispectral Index (BIS) using non-invasive device. At values near 100 mean patient is more likely to be awake and at values below 60 are more likely to be under general anesthesia.
Bispectral Index after 8 minutes | 8 minutes after general anesthesia induction
  Bispectral Index (BIS) using non-invasive device. At values near 100 mean patient is more likely to be awake and at values below 60 are more likely to be under general anesthesia.
Bispectral Index after 10 minutes | 10 minutes after general anesthesia induction
  Bispectral Index (BIS) using non-invasive device. At values near 100 mean patient is more likely to be awake and at values below 60 are more likely to be under general anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel MN Guimaraes, MSc, Principal Investigator — Professor
Locations (1):
- Hospital Universitário de Brasilia, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Plan to share at open database.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: After study ends
Access Criteria: Open